CLINICAL TRIAL: NCT05253001
Title: Effects of Antenatal Education on Maternal Childbirth Self-efficacy and Satisfaction
Brief Title: Effects of Antenatal Education on Maternal Childbirth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Ching-Yi Chang, Department of School of Nursing, Taipei Medical University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: TMU109-AE1-B25
Record Dates: First submitted 2022-01-05; First posted 2022-02-23 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Self Efficacy; Maternal Behavior
Keywords: maternal self-efficacy; maternal education

STUDY DESIGN:
Intervention Model Description: An experiment was developed in the current study. A total of 40 women from a medical hospital in northern Taiwan were recruited as the participants. The study groups mobile chatbot approach to improving prenatal education. The controp group was a traditional approach to prenatal education.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): use mobile chatbot approach to improve prenatal education
  Interventions: Device: smartphone
- controp group (Placebo Comparator): a traditional approach to prenatal education
  Interventions: Device: smartphone

INTERVENTIONS:
Device: smartphone — Use the mobile chatbot approach for intervention groups to improve prenatal education.

SUMMARY:
In prenatal education, pregnant women's knowledge is a crucial issue for protecting pregnant women and newborns healthy. Therefore, prenatal education has become a basic and essential program for each pregnant woman. However, most of the current prenatal education courses are taught via a group teaching approach, which makes it difficult for pregnant women to think deeply about relevant birth issues due to the lack of interaction and context. This may in turn have an impact on childbirth choice and clinical judgment.

DETAILED DESCRIPTION:
My study Purpose wants to see doseThe mobile chatbot approach improve prenatal education shared decision-making. In order to verify the effectiveness of such a learning design, an experiment was developed in the current study. A total of 40 women from a medical hospital in northern Taiwan were recruited as the participants.

ELIGIBILITY:
Inclusion Criteria:

* Parturients who have come to the hospital for obstetrics

Exclusion Criteria:

* Parturients who have ever to the hospital for obstetrics

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Effects of antenatal education on maternal childbirth self-efficacy and satisfaction | the outcome measure will be assessed through study completion and data will be reported up to 1 year.
  The study will be using the maternal childbirth self-efficacy questionnaire to survey the participants' use outcomes related the smartphone use.
Effects of antenatal education on maternal childbirth self-efficacy and satisfaction | the outcome measure will be assessed through study completion and data will be reported up to 1 year.
  The study will use the maternal childbirth satisfaction questionnaire to survey the participants' childbirth experience related to smartphone use.

IPD SHARING:
Plan to Share IPD: No